CLINICAL TRIAL: NCT01217333
Title: Telephone-Based Decision Support for Rural Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Breast Cancer Research Program (Other)
Responsible Party: Principal Investigator, Jeff Belkora, Assistant Professor, Surgery and Health Policy Director, Decision Services, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CBCRP 12BB-3900
Record Dates: First submitted 2010-09-28; First posted 2010-10-08 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Breast Cancer
Keywords: Telephones; Community-Based Participatory Research; Participation, Patient; Rural health services
MeSH Terms: conditions — Breast Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-person (Active Comparator): Participants in this arm have been randomized to receive Consultation Planning in-person
  Interventions: Behavioral: In-person CP
- Telephone (Active Comparator): Participants in this arm have been randomized to receive Consultation Planning by telephone.
  Interventions: Behavioral: Tele-CP

INTERVENTIONS:
Behavioral: In-person CP — CP is a structured interview in which a lay health worker prompts a patient to articulate questions and concerns about decision issues in preparation for a treatment discussion with a provider. The Consultation Planner (CPer) then completes and prints out a word-processed template, paraphrasing and summarizing the patient's questions and concerns. The patient takes away the printed Consultation Plan to serve as a visual aid and agenda during the meeting with the doctor. CPers are trained to avoid providing medical advice or information. Arrangements will be made for participants who do not have transportation to the CRCMC.
  Other Names: SCOPED Model; Question listing
  Arms: In-person
Behavioral: Tele-CP — Participants in the Tele-CP arm will receive CP by telephone. Arrangements will be made for participants who do not have access to a telephone.
  Other Names: SCOPED Model; Question listing
  Arms: Telephone

SUMMARY:
The investigators community based resource center has implemented visit preparation by prompting patients to write down their questions. This is a proven approach to increasing the number of questions and concerns that patients voice during their visits with doctors. The resource center's usual practice is to provide their visit preparation intervention, called Consultation Planning, through in-person counseling sessions. This study asks whether telephone delivery of Consultation Planning would be almost as effective in terms of increasing patient's decision self-efficacy, or confidence in their ability to navigate decisions effectively with their physicians. The study also asks about the cost-effectiveness of telephone delivery compared to in-person delivery. The investigators are answering these questions through a randomized, controlled, non-inferiority trial with two arms: in-person versus telephone delivery of Consultation Planning. The investigators are measuring self-reported psychological outcomes such as decision self-efficacy (primary outcome), preparation for decision making, anxiety, and distress, along with economic outcomes such as health resource utilization and willingness to pay. The investigators hypothesize that Tele-CP can be delivered at a lower patient and resource center cost than in-person CP, and that it will be as effective in terms of impact on a patient's decisional self-efficacy.

DETAILED DESCRIPTION:
Breast cancer patients are often advised to write down a list of questions before talking to their surgeons or oncologists about treatment decisions. However, without support, newly diagnosed patients may be too overwhelmed to make a list of their questions. Over the last 30 years, studies have shown that patients benefit from having a researcher or nurse prompt them for questions or any concerns they may have before an upcoming appointment with their primary healthcare provider. In some of these studies, the researcher or nurse then wrote down the patient's questions so that the clinician could be sure to address them.

Today, few facilities provide this type of patient support, known as visit preparation, perhaps because of the cost and/or organizational challenges. Our research team, a partnership between the UCSF Decision Services and the Cancer Resource Centers of Mendocino County (CRCMC) implemented a form of visit preparation known as Consultation Planning (CP). The investigators have made CP work in our communities by training resource center staff to deliver the service in face-to-face interviews with patients.

In a recent completed Pilot Study, the investigators collected and analyzed initial data suggesting that CP is appropriate for diverse, rural patients in Mendocino County (including Native Americans and Latinas), and that CP may be effective when delivered by telephone.

The investigators have now been awarded a grant to examine the effectiveness and cost-effectiveness of delivering CP by telephone (Tele-CP) versus in person.

Primary Objectives:

* To measure and compare the impact of in-person CP and Tele-CP on decisional self-efficacy (primary outcome), decisional conflict, anxiety, breast cancer-related quality of life, and adherence to visits and treatments.
* To measure and compare the cost-effectiveness of in-person CP and Tele-CP

Secondary Objective:

• To measure physician satisfaction and perception of the decision process.

Study Hypotheses:

1. Tele-CP can be delivered at a lower patient and resource center intervention cost than in-person CP.
2. Tele-CP patients will reach the same levels of decisional self-efficacy (primary outcome), decisional conflict, anxiety, quality of life, and adherence to visits and treatment as in-person CP patients.
3. Physicians will report equal satisfaction and will rate their decision process equally whether the patient experienced CP or Tele-CP.

In 1996, Dr. Belkora and his colleagues evaluated CP at Stanford and UCSF, finding that it reduced perceived barriers to communication and improved satisfaction for patients and physicians. CP has been available at the UCSF Cancer Resource Center since 1999, where it is advertised to all cancer patients through brochures and flyers. CP has also been integrated into the clinical processes at the UCSF Breast Care Center since 1998, where it is now offered to every patient with new or locally recurrent disease who is facing early-stage breast cancer treatment decisions.

In 2003, Dr. Belkora was awarded research funding from the California Breast Cancer Research Program to implement a Pilot Study entitled: Decision Support in Rural Underserved North Coast Counties. This pilot project documented, in a retrospective design, that both onsite and Tele-CP were associated with high satisfaction or decision self-efficacy levels among rural cancer patients who received non-medical supportive services from the CRCMC.

The investigators therefore concluded that CP and Tele-CP are acceptable, feasible, and viable interventions to compare in a prospective randomized, controlled trial in Mendocino County. The investigators were also able to conclude that the Decision Self Efficacy was a suitable primary outcome measure from both the scientific and community viewpoints.

This study is a non-inferiority design which is used in situations where an effective treatment has already been established, in this case in-person CP. The goal is to prove, statistically, that another treatment (Tele-CP) is as effective as the established one, within a predetermined margin of non-inferiority. We will therefore conduct a randomized, controlled trial of non-inferiority between Tele-CP and in-person CP. The outcomes include decisional self-efficacy, anxiety, decisional conflict, disease-related quality of life, adherence to visits and treatments, intervention costs to the patient and resource center as well as physician satisfaction and perception of the decision process.

Approximately 90 Mendocino patients are diagnosed every year with new or locally recurrent breast cancer. An average of 75 breast cancer patients per year become clients of the CRCMC, in that they receive non-medical supportive services from this agency. For example, resource center clients are matched with a "buddy" who is a survivor of a similar condition and is trained to provide emotional support. Clients also use the resource center library and attend support groups. In the past, they have been offered in-person CP.

Once our study begins, all resource center clients diagnosed with stage 0, 1, 2, 3, or 4 breast cancer and who are scheduled for a decision making appointment with a surgeon or oncologist will be asked to participate. Based on updated preliminary data (from the resource center's 2007 records), the investigators will require 58 subjects over the study period in order to make the primary analysis of the study scientifically and statistically valid, although we will continuing accruing up to 116 patients in order to conduct secondary, exploratory, subset analyses. Clients who consent to participate in our study will be randomly assigned to Tele-CP or in-person CP. A resource center staff member (Consultation Planner or "CPer") will use the assigned method (CP or Tele-CP) to help the patients prepare a list of questions for their surgeon or oncologist. Before and after the CP or Tele-CP session and their doctor's appointment, clients will be asked to complete short surveys describing their confidence, anxiety, confusion, quality of life, and costs to them of doing the CP session (e.g. travel time). From these surveys, as well as other records, we will determine whether Tele-CP is as effective as in-person CP, and whether it was more convenient and less costly.

Time 0:

* When a patient with breast cancer contacts CRCMC for information or support, the CRCMC staff will ask the client to complete the standard CRCMC Client Intake Form. Staff will then offer CP and inquire about the client's potential interest in participating in the study. If the client is a monolingual Spanish speaker, the resource center staff will enlist one of the designated translators to assist with the communication and consent process, utilizing our UCSF CHR approved Spanish Consent Form. If the client has any potential interest in study participation, she will then be referred to a member of the research team. The client will also be given a copy of the UCSF CHR approved study consent form for their review.
* A member of the research team will review the study protocol with the CRCMC client and proceed with the informed consent process.
* For frontier clients (living in extremely remote areas), the consent process will be initiated on the phone with a member of the research team, and a copy of the consent form will be mailed, faxed, or emailed to the subject. After the subject has had a chance to read and review the consent, the research team member will then address (via telephone) all questions or concerns they may have. If the subject wishes to proceed with the study, she will then sign the consent and forward it back to the research team member by fax or US mail.
* For subjects who can easily be met in person and do not have transportation challenges, a research team member will meet with each subject and complete the consent process in person.

Each consent process will be completed pursuant to all UCSF, State and Federal Guidelines for the Protection of Human Subjects. No study procedures will be initiated until after the consent process is complete and the subject signs the study consent form. A copy of the consent will be given to each subject. A copy of these documents will also be placed in the subject's CRCMC client file.

This trial will take place at the inland and coastal offices of the CRCMC located in Ukiah and Mendocino. Interventions will take place by telephone in one study arm, and at a resource center office site (Ukiah or Mendocino, depending on which is closer to the client domicile) in the other study arm. Patients randomized to the resource center arm, who cannot arrange for transport, will be driven by a resource center staff member.

Time 1:

• After an informed consent is obtained, a research team member will then initiate the study protocol procedures, obtain random assignment and schedule the patient for the appropriate CP intervention.

Time 2:

• The Consultation Planner (CPer, i.e. study interventionist) will meet with the client (and translators if necessary) either at the resource center or over the telephone via conference call. The CPer will administer the baseline surveys in-person or by phone, then the CPer will administer CP, and finally, once the participant has received a printed copy of the CP, the CPer will administer post-CP surveys. The CPer will audiorecord this session whether it takes place in person or by telephone. Participants who receive Tele-CP will receive a copy of the printed CP either by mail, fax, email, or in-person. Consistent with resource center practices, during the Tele-CP call the CPer will arrange a mutually convenient time to meet with the participant either by phone or in person to review the printed CP. The Post-CP surveys will be administered at this time.

Time 3:

* The CPer, (and translator if necessary) will accompany the patient to her doctor's appointment with the specialist. The CPer will audiorecord the visit (patients will be mailed a copy of the audiorecording within a week), and administer post-visit surveys immediately at the conclusion of the appointment. The subjects will also receive a copy of the CPer notes for their review and files.
* Because the investigators are incorporating a survey for clinicians to complete after the consultation, the investigators have also included a Physician Consent Form for the study. A research team member will also provide to each participating clinician a copy of the study consent form and review the study with each of these subjects. An informed consent will be completed with each clinician. A copy of the consent (including the Experimental Subject's Bill of Rights) will be given to each physician. At the start of the study, the investigators will approach all Mendocino oncologists and surgeons who see breast cancer patients to determine their willingness to participate.
* Note: This Physician consent process will be completed pursuant to all UCSF, State and Federal Guidelines for the Protection of Human Subjects. No study procedures will be initiated until after the consent process is complete and the physician signs the study consent form. A copy of the consent (including the Experimental Subject's Bill of Rights) will be given to these subjects.

Time 4:

Six months following the physician consultation, the a research team member will contact the client (and translator if needed) to complete the 6 month surveys. At this time, a copy of the participant's current CRCMC Client Intake form will be added to the study file.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18 or older
* Diagnosis of Ductal Carcinoma in Situ (DCIS) or local recurrence of DCIS
* New (stage 1, 2, 3, 4) invasive breast cancer or recurrence
* Upcoming appointment to see a surgeon or oncologist to discuss treatment options
* Surgeons or oncologists whom the patient is consulting
* Able to speak, read, and understand English or Spanish

Exclusion Criteria:

* Females less than 18 years of age
* Males with breast cancer
* Females with breast cancer who are also pregnant (pregnancy changes the breast cancer treatment)
* Clients who are determined to have "diminished mental capacity" according to the standards of the CRCMC Policy on Mental Competence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Decisional Self-Efficacy (DSE) | -1 hour (1 hour prior to intervention)
Decisional Self-Efficacy (DSE) | 5 min after intervention

SECONDARY OUTCOMES:
CRCMC Client Intake Form | Immediately upon consent
STAI Form Y-1 (Anxiety) | -1 hour (1 hour prior to intervention)
Decisional Conflict Scale (DCS) | -1 hour (1 hour prior to intervention)
Critical Incident Survey | 5 min (5 minutes after intervention)
Patient Intervention Costs | 5 min (5 minutes after intervention)
Patient Utility Assessments | 5 min (5 minutes after intervention)
Quality of Life Thermometer | Immediately upon consent
Preparation for Decision Making (PDM) Scale | 5 min (5 minutes after intervention)
Tracking Log of Medical Visits and Treatments | 1 week avg. (immediately following appointment with specialist)
Patient Healthcare Costs | Immediately upon consent; 6 months after intervention
STAI Y-1 (Anxiety) | 5 minutes after intervention
Decisional Conflict Scale (DCS) | 1 week avg. (immediately following visit with physician)
Critical Incident Survey | 1 week avg. (immediately following visit with physician)
Patient Intervention Costs | 1 week avg. (immediately following visit with physician)
Patient Utility Assessments | 6 months after intervention
Quality of Life Thermometer | 6 months after intervention
Preparation for Decision Making (PDM) Scale | 6 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Belkora, Ph.D., Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Cancer Resource Centers of Mendocino County, Mendocino, California
  - Cancer Resource Centers of Mendocino County, Ukiah, California

REFERENCES:
- [Result] Belkora J, Stupar L, O'Donnell S, Loucks A, Moore D, Jupiter C, Johnson N, Wilson L. Decision support by telephone: randomized controlled trial in a rural community setting. Patient Educ Couns. 2012 Oct;89(1):134-42. doi: 10.1016/j.pec.2012.06.009. Epub 2012 Jul 7. PMID 22776761